CLINICAL TRIAL: NCT05149131
Title: A reAl-World Evidence Study Using Alberta Population Based Data to Describe Treatment Patterns for Metastatic castRation sENsitivE proState Cancer patientS (AWARENESS)
Brief Title: A Study Called AWARENESS Using Data From Men in Alberta to Observe Treatment Patterns for Metastatic Castration-sensitive Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21991
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Castration-sensitive Prostate Cancer
MeSH Terms: interventions — Androgen Antagonists; luprolide acetate gel depot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mCSPC patients in the province of Alberta: mCSPC patients who initiated and received at least one dose of guideline recommended life-prolonging therapy for mCSPC (docetaxel, abiraterone, enzalutamide, apalutamide, or ADT alone) from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff, inclusive.
  Interventions: Drug: ADT (Eligard®*) with or without treatment intensification

INTERVENTIONS:
Drug: ADT (Eligard®*) with or without treatment intensification — Abiraterone acetate (Zytiga®) Enzalutamide (Xtandi®) Apalutamide (Erleada®) Docetaxel (Taxotere®)
  *may be substituted with leuroprolide gel, buserelin, goserelin, triptorelin, histrelin, cyproterone or degarelix

SUMMARY:
This is an observational study in which patient data from the past on men with metastatic castration-sensitive prostate cancer is studied.

Metastatic castration-sensitive prostate cancer (mCSPC) is a type of advanced prostate cancer that has spread to other parts of the body, and still responds to treatment that lowers testosterone levels.

Cancer is a condition in which the body cannot control the growth of cells. The extra cells can form tumors in organs or other parts of the body. If tumors form in the prostate, male hormones (androgens) can sometimes help the cancer spread and grow. The main hormone that does this is called testosterone and is mainly made in the testicles. Men with prostate cancer can have treatments to try to lower the levels of testosterone in the body. One possible treatment is surgery to remove the testicles. Another option is taking treatments to lower the levels of testosterone in the body. These are called androgen deprivation therapy (ADT). In men with mCSPC, ADT can help to stop the cancer from growing and spreading. Men with mCSPC can also receive "treatment intensification". This means that they receive ADT as well as other treatments for their prostate cancer. Other studies that looked at treatment of mCSPC in Canada have found that most men with mCSPC do not receive treatment intensification.

In this study, the researchers want to collect more data about the men who had mCSPC and the types of treatment they received for their mCSPC. The researchers will look at the health information of adult men in Alberta, Canada who had at least 1 dose of treatment for their mCSPC between January 2016 and December 2020 or earlier.

The study will first look at the health information of men whose cancer had metastasized or spread to other parts of the body, beyond the prostate, at the time they were diagnosed with prostate cancer.

And later, if feasible to do, the study may also look at the health information from men who were diagnosed with prostate cancer that was limited to the prostate, and over time spread to other parts of the body.

The researchers will collect information from databases, a census, and pharmacy records. This will help the researchers learn more about:

* whether the men received ADT alone, or ADT with treatment intensification
* additional information about the men, including their age, income, level of education, residential area (urban or rural) and the more information about the treatments received
* how the men's symptoms affected their daily lives
* how severe the men's cancer was
* changes in laboratory values as markers for changes to the blood, liver, kidney, bone or other organs
* need for additional treatment
* where the men's cancer may have spread to in other parts of the body.

There will be no required visits with a study doctor or required tests in this study since it's reviewing patient data from the past.

The researchers will collect this information for about 7 months. The entire study will take about 10 months to finish.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Diagnosed with mCSPC
* Residents of Alberta, Canada
* Initiating ADT with or without treatment intensification from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff

Exclusion Criteria:

- There are no formal exclusion criteria in order to capture real-world utilization of ADT with or without treatment intensification

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all mCSPC patients in the province of Alberta that initiated and received at least one dose of guideline recommended life-prolonging therapy for mCSPC (docetaxel, abiraterone, enzalutamide, apalutamide, or ADT alone) from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff, inclusive.
  Patients with de novo metastatic disease are easily identifiable by diagnosis with metastatic disease. Patients who relapse with metastatic disease may be more challenging to identify. The study will start by reporting on results for de novo mCSPC patients only while feasibility assessment is done to determine if these patients can be identified, and if so, they will be added to the study population.
Sampling Method: Non-Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of patient characteristics by cohort | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff

SECONDARY OUTCOMES:
Change in percentage of patients within each treatment cohort by year | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Overall survival | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Percentage of patients that died due to cancer | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Percentage of patients that received subsequent life-prolonging therapies (LPT) | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Attrition rate for each line of therapy | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Total incidence (number) of hospitalizations | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff
Total incidence (number) of emergency department visits | Retrospective analysis from 01-Jan-2016 up to 31-Dec-2020 or earlier based on database cutoff

CONTACTS AND LOCATIONS:
Locations (1):
- Databases, Multiple Locations, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.